CLINICAL TRIAL: NCT02804893
Title: Prospective, Randomized, Multicentric Study On Videothoracoscopic (Vats) Vs Robotic Approach For Lobectomy Or Anatomical Segmentectomy In Patients Affected By Early Lung Cancer (ROMAN)
Brief Title: Videothoracoscopic (VATS) vs. Robotic Approach for Lobectomy or Anatomical Segmentectomy
Acronym: ROMAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Fondazione Umberto Veronesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1566
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Lung Cancer
Keywords: Lung cancer, video-assisted thoracoscopic surgery, robotic-assisted thoracoscopic surgery
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VATS GROUP (Active Comparator): VATS lobectomy or segmentectomy
  Interventions: Procedure: VATS
- RATS GROUP (Active Comparator): Robotic lobectomy or segmentectomy
  Interventions: Procedure: RATS

INTERVENTIONS:
Procedure: VATS — Thorax thoracoscopic surgery (lobectomy)
  Other Names: Minimally invasive video-assisted surgery
  Arms: VATS GROUP
Procedure: RATS — Thorax robotic surgery (lobectomy)
  Other Names: Minimally invasive robot-assisted surgery
  Arms: RATS GROUP

SUMMARY:
This is a prospective, randomized, multicenter study on 300 patients (150 VATS lobectomies and 150 robotic lobectomies) affected by early stage (I-II) lung cancer. The expected recruitment is one year and two year follow up. Surgeons should have a minimum of 30 major lung resections performed using one of the two techniques for participation in the study. Each participating centers should have the possibility to offer both techniques (Robotics and Vats). The primary end point is a combination of conversion and complication rate. The presence of at least one of the two events is considered a failure. Considering the rate of failure of 35% in the VATS arm, we want to see a failure rate not over 20% in the robot arm, so with a power of 80% and an alpha error of 5%, we need a total of 300 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old
* Known or suspected lung cancers
* Patients in clinical stage T1-T2, N0-N1 candidate to surgery lobectomy or anatomical segmentectomy
* ASA-1-2-3

Exclusion Criteria:

* Clinical stage >II
* Severe heart disease
* Alcohol abuse
* Renal impairment (creatinine >2.5)
* Presence of serious comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-03-06 (Estimated); Study Completion 2023-03-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative complications: conversion rate, defined as procedures that start with minimally invasive access and are converted to open surgery due to different reasons (bleeding, anatomical reasons, oncological reasons, technical reasons, other) | date of Surgery
Postoperative complications: surgical complications, higher or equal grade II assessed by Clavien-Dindo scale, within 90 days | within 90 days

SECONDARY OUTCOMES:
Duration of surgery | date of Surgery
Number of resected lymph nodes and upstaging | date of Surgery
Proportion of patients who undergo complete resection during the procedure | date of Surgery
Postoperative hospital stay | 2 weeks
Postoperative pain: daily evaluation with visual numeric scale before and after surgery until discharge | 2 weeks, 6 months and 12 months
Quality of life by EORTC QOL-C30 | 2 weeks, 6 months and 12 months
Duration of analgesic use after discharge and time to return to normal daily activity | within 90 days
Postoperative respiratory function: FEV 1, PEF and CV | 6 month postoperatively
Rate of local and distant recurrence and disease free survival | 24 months
Patient's immune response: analysis of PCR, serum interleukins, lymphocytes subpopulations | before surgery, 2 hours after surgery and at 3rd and 14th postoperative day

CONTACTS AND LOCATIONS:
Locations (1):
- Thoracic surgery Division, Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Demmy TL, Curtis JJ. Minimally invasive lobectomy directed toward frail and high-risk patients: a case-control study. Ann Thorac Surg. 1999 Jul;68(1):194-200. doi: 10.1016/s0003-4975(99)00467-1. PMID 10421140
- [Result] Hoksch B, Ablassmaier B, Walter M, Muller JM. [Complication rate after thoracoscopic and conventional lobectomy]. Zentralbl Chir. 2003 Feb;128(2):106-10. doi: 10.1055/s-2003-37763. German. PMID 12632277
- [Result] Nakata M, Saeki H, Yokoyama N, Kurita A, Takiyama W, Takashima S. Pulmonary function after lobectomy: video-assisted thoracic surgery versus thoracotomy. Ann Thorac Surg. 2000 Sep;70(3):938-41. doi: 10.1016/s0003-4975(00)01513-7. PMID 11016337
- [Result] Nomori H, Ohtsuka T, Horio H, Naruke T, Suemasu K. Difference in the impairment of vital capacity and 6-minute walking after a lobectomy performed by thoracoscopic surgery, an anterior limited thoracotomy, an anteroaxillary thoracotomy, and a posterolateral thoracotomy. Surg Today. 2003;33(1):7-12. doi: 10.1007/s005950300001. PMID 12560900
- [Result] Yim AP, Wan S, Lee TW, Arifi AA. VATS lobectomy reduces cytokine responses compared with conventional surgery. Ann Thorac Surg. 2000 Jul;70(1):243-7. doi: 10.1016/s0003-4975(00)01258-3. PMID 10921716
- [Result] Li WW, Lee RL, Lee TW, Ng CS, Sihoe AD, Wan IY, Arifi AA, Yim AP. The impact of thoracic surgical access on early shoulder function: video-assisted thoracic surgery versus posterolateral thoracotomy. Eur J Cardiothorac Surg. 2003 Mar;23(3):390-6. doi: 10.1016/s1010-7940(02)00795-9. PMID 12614812
- [Result] McKenna RJ Jr, Wolf RK, Brenner M, Fischel RJ, Wurnig P. Is lobectomy by video-assisted thoracic surgery an adequate cancer operation? Ann Thorac Surg. 1998 Dec;66(6):1903-8. doi: 10.1016/s0003-4975(98)01166-7. PMID 9930466
- [Result] Leschber G, Holinka G, Linder A. Video-assisted mediastinoscopic lymphadenectomy (VAMLA)--a method for systematic mediastinal lymphnode dissection. Eur J Cardiothorac Surg. 2003 Aug;24(2):192-5. doi: 10.1016/s1010-7940(03)00253-7. PMID 12895606
- [Result] Yim AP, Landreneau RJ, Izzat MB, Fung AL, Wan S. Is video-assisted thoracoscopic lobectomy a unified approach? Ann Thorac Surg. 1998 Oct;66(4):1155-8. doi: 10.1016/s0003-4975(98)00622-5. PMID 9800798
- [Result] Cao C, Tian DH, Wolak K, Oparka J, He J, Dunning J, Walker WS, Yan TD. Cross-sectional survey on lobectomy approach (X-SOLA). Chest. 2014 Aug;146(2):292-298. doi: 10.1378/chest.13-1075. PMID 24504007
- [Result] Daniels LJ, Balderson SS, Onaitis MW, D'Amico TA. Thoracoscopic lobectomy: a safe and effective strategy for patients with stage I lung cancer. Ann Thorac Surg. 2002 Sep;74(3):860-4. doi: 10.1016/s0003-4975(02)03764-5. PMID 12238851
- [Result] Melfi FM, Menconi GF, Mariani AM, Angeletti CA. Early experience with robotic technology for thoracoscopic surgery. Eur J Cardiothorac Surg. 2002 May;21(5):864-8. doi: 10.1016/s1010-7940(02)00102-1. PMID 12062276
- [Result] Park BJ, Flores RM, Rusch VW. Robotic assistance for video-assisted thoracic surgical lobectomy: technique and initial results. J Thorac Cardiovasc Surg. 2006 Jan;131(1):54-9. doi: 10.1016/j.jtcvs.2005.07.031. PMID 16399294
- [Result] Gharagozloo F, Margolis M, Tempesta B, Strother E, Najam F. Robot-assisted lobectomy for early-stage lung cancer: report of 100 consecutive cases. Ann Thorac Surg. 2009 Aug;88(2):380-4. doi: 10.1016/j.athoracsur.2009.04.039. PMID 19632377
- [Result] Veronesi G, Galetta D, Maisonneuve P, Melfi F, Schmid RA, Borri A, Vannucci F, Spaggiari L. Four-arm robotic lobectomy for the treatment of early-stage lung cancer. J Thorac Cardiovasc Surg. 2010 Jul;140(1):19-25. doi: 10.1016/j.jtcvs.2009.10.025. Epub 2009 Dec 28. PMID 20038475
- [Result] Louie BE, Farivar AS, Aye RW, Vallieres E. Early experience with robotic lung resection results in similar operative outcomes and morbidity when compared with matched video-assisted thoracoscopic surgery cases. Ann Thorac Surg. 2012 May;93(5):1598-604; discussion 1604-5. doi: 10.1016/j.athoracsur.2012.01.067. Epub 2012 Mar 20. PMID 22440364
- [Result] Nakamura H. Systematic review of published studies on safety and efficacy of thoracoscopic and robot-assisted lobectomy for lung cancer. Ann Thorac Cardiovasc Surg. 2014;20(2):93-8. doi: 10.5761/atcs.ra.13-00314. Epub 2014 Feb 28. PMID 24583699
- [Derived] Veronesi G, Abbas AE, Muriana P, Lembo R, Bottoni E, Perroni G, Testori A, Dieci E, Bakhos CT, Car S, Luzzi L, Alloisio M, Novellis P. Perioperative Outcome of Robotic Approach Versus Manual Videothoracoscopic Major Resection in Patients Affected by Early Lung Cancer: Results of a Randomized Multicentric Study (ROMAN Study). Front Oncol. 2021 Sep 9;11:726408. doi: 10.3389/fonc.2021.726408. eCollection 2021. PMID 34568057